CLINICAL TRIAL: NCT06527053
Title: Evaluation of Digital Versus Conventional Roofless Obturators in Partial Maxillectomy Cases
Brief Title: Digital Obturators in Maxillectomy Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Nasr, Assistant Lecturer Eman Nasr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RP08-21\4
Record Dates: First submitted 2024-04-15; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Device Malfunction
Keywords: digital obturators-roofless design-maxillectomy-mucorycosis

STUDY DESIGN:
Intervention Model Description: patients with maxillary defects had received two types of obturators
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- digital obturator (Experimental): new approach to create device
  Interventions: Device: obturator
- conventional obturator (Experimental): old approach to create device
  Interventions: Device: obturator

INTERVENTIONS:
Device: obturator — special maxillofacial device to close hollow defects

SUMMARY:
Using Digital approach to treat patients with maxillofacial defects without surgical intervention

DETAILED DESCRIPTION:
Evaluating digital dental and maxillofacial obturators to artifitially close maxillofacial defects in paients with oral cancer and patients with mucormycosis fungal post covid infection.

Craeting Digitized database for all patients included in the study.

Recording casses with post covid infection in specific period.

ELIGIBILITY:
Inclusion Criteria:

-

All participants in this study will be selected according to the following criteria:

* Patients with maxillary defects Class I and class II Aramany Classification with completely healed tissues.
* Patients' age ranging from 20 to 70 years old.
* Nearly intact mandibular arch.

Exclusion Criteria:

-

Participants with the following criteria will be excluded from the study:

* Physical or mental instability.
* Completely edentulous patients.
* Patients presenting allergy to materials being used.
* Patients lacking compliance to maintain acceptable oral hygiene.
* Patients taking radiotherapy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of hypernasality in speech | one month
  physiologic parameter
Evaluation of masseter muscle muscle | three months
  physiologic parameter
Evaluation of Patient Quality of Life | six months
  questionnaire
Evaluation of retention | 1 day (at time of device insertion)
  descriptive by KP scale
Obturator misfit | 1 day (at time of device delivery)
  descriptive by Digital software

CONTACTS AND LOCATIONS:
Overall Officials: ali al shaikh, professor, Principal Investigator — Tanta University
Locations (1):
- Eman Nasr, Tanta, Gharbia Governorate, Egypt